CLINICAL TRIAL: NCT03709667
Title: Exercise in Methamphetamine Use Disorder: Dopamine Receptor Upregulation and Neural Function
Brief Title: Exercise in Methamphetamine Use Disorder Upregulation and Neural Function
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Edythe London, Professor of Psychiatry and Biobehavioral Sciences and Molecular and Medical Pharmacology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-000496; R01DA045162 (NIH)
Record Dates: First submitted 2018-07-12; First posted 2018-10-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Methamphetamine Abuse
Keywords: exercise; methamphetamine
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EX (Experimental): Participants in this arm of the study will be randomized in to the exercise intervention.
  Interventions: Behavioral: EX
- CON (Placebo Comparator): The control condition is a health-education intervention.
  Interventions: Behavioral: CON

INTERVENTIONS:
Behavioral: EX — An individualized aerobic and resistance-exercise program will be developed for each participant on the basis of a maximal incremental exercise test and strength assessments performed at baseline. This test will measure aerobic capacity (VO2 max) and the metabolic or lactate threshold (VO2θ) (i.e., the level of O2 uptake that defines one's ability to perform prolonged work), using indirect calorimetry with an automated metabolic-measurement system. The intervention will comprise 24 sessions over 8 wk (3x/wk), supervised by a credentialed exercise specialist. Each session will consist of a 5-min warm-up, 30-40 min of aerobic activity on a treadmill, 15-20 min of resistance training, and a 5-min cool-down.
  Arms: EX
Behavioral: CON — Participants attend 50-min sessions 3x/wk matched to EX for staff contact. A counselor will facilitate integrative group discussions, and will conduct a multimedia program addressing various health, wellness and lifestyle topics, such as nutrition, dental care, stress relief, sleep hygiene, relationships, immunizations, health screening, smoking, environmental health, and time management.
  Arms: CON

SUMMARY:
The purpose of this research study is to determine the effects of an exercise intervention and health-education program on brain dopamine receptors and on cognitive functions that have been linked to these receptors.

DETAILED DESCRIPTION:
After completing baseline assessments within 2 wks after admission, participants will be randomized to one of two interventions: Exercise (EX, active intervention), consisting of 3x-weekly 50-min aerobic + resistance-training sessions for 8 wk; Health Education (control intervention, CON), consisting of 50-min health education sessions 3x-weekly for 8 wk. Participants will undergo positron emission tomography (PET) and functional magnetic resonance imaging (fMRI) scans while performing the stop signal task (SST) and the reversal learning task (RLT) (cognitive computer tasks) at baseline and after completing the 8-wk protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Language: Participants must be fluent in English, as demonstrated by verbal skills sufficient to participate in a conversation, including the ability to ask and answer questions at a level that assures adequate understanding of the study. A comprehension quiz will be administered.
2. Age 18-65 years
3. Meets Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for moderate to severe stimulant use disorder assessed by MINI.
4. Vital Signs: Within the clinically acceptable normal range (e.g., resting pulse 50 to 99/min, blood pressure between 85-150 mm Hg systolic and 45-90 mm Hg diastolic.
5. Labs: hematology and chemistry laboratory test results within normal (+/- 10%) limits.
6. Right handed.

Exclusion Criteria:

1. Neurological disease: history of seizure disorder, brain injury with loss of consciousness > 30 min, or other neurological disorder that would interfere with informed consent, data interpretation or participant safety.
2. Musculoskeletal disease that would prevent participation in exercise.
3. Current psychotic disorder assessed by the MINI.
4. Current suicidal ideation/plan, assessed by the Patient Health Questionnaire-9.
5. Heart disease: Hypertension or unstable pulmonary or cardiovascular disease that would interfere with participation in the EX regimen
6. Evidence of untreated or unstable medical illness, including endocrine, autoimmune, renal, hepatic, or active infectious disease, which might compromise safe participation (HIV+ participants must be receiving a stable regimen of antiretroviral medication throughout the course of the study).
7. Pregnancy [Women must provide negative pregnancy urine tests before study entry].
8. Asthma or use of theophylline, α- and β-adrenergic agonists, or other sympathomimetics.
9. Medications: Antihypertensive agents, antidepressants, and antiretroviral medications are prescribed to some clients at Cri-Help. Any participant taking any medication that has direct dopaminergic action (e.g., bupropion, neuroleptics) will be excluded, but other chronic medications such as selective serotonin reuptake inhibitors will be allowed. Any participant taking a medication chronically must maintain a stable dose throughout the study; antiretrovirals and antidepressants must be initiated at least 1 week before baseline scan.
10. Radiation Exposure: Participants who have participated in any other research study involving exposure to ionizing radiation in the past year if the total cumulative dose from the past research studies and the current research study would exceed the limits described by the FDA in 21 Code of Federal Regulations 361.1. Specifically, the total annual cumulative dose to the body, active blood-forming organs, lens of the eye and gonads must remain below 5 rems and the total annual cumulative dose to all other organs must remain below 15 rems. Potential participants who have had exposure to ionizing radiation in the past year cannot be allowed to participate if the investigators are unable to obtain proper documentation quantifying the amount of past exposure.
11. Metal devices: (e.g., pacemaker, infusion pump, aneurysm clip, prosthesis, plate) in the body.Presence of such a device could interfere with scan acquisition or pose a potential risk during MRI. [A participant who has an implanted device can enroll with documentation that the device is MRI-compatible.
12. Claustrophobia: Subjects will be questioned about their potential discomfort with enclosed spaces, such as an MRI scanner. Subjects reporting problems with enclosed spaces will be excluded.
13. Any other condition that would compromise safe participation, determined by the study physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Striatal D2/3 Binding Potential (BPND) Upregulation | 8 weeks
  Dopamine D2-type receptor binding potential in the striatum measured with positron emission tomography scanning measured at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment.

SECONDARY OUTCOMES:
Sustained attention | 8 weeks
  The Continuous Performance Task will be used to assess sustained attention at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment. The following outcome variables will be assessed:
  Correct Detection: Number of responses to the target stimulus. Reaction times: Length of time between stimulus presentation and response. Omission errors: Number of target presentations with no response. Commission errors: Number of responses without target stimulus presentation.
  High omission rates reflect impaired attention, higher correct detections reflect improved attention.
Working memory | 8 weeks
  The Sternberg Spatial Task will be used to assess working memory at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment. The number of correct responses will be measured, with higher amounts of correct responses reflecting better working memory.
Declarative memory | 8 weeks
  The Rey Auditory Verbal Learning Test will be used to assess declarative memory at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment. The number of words correctly recalled will be recorded before and after a 20 minute delay, as well as the number of intrusions. The corresponding Z score and percentile of each participant's responses will be calculated.
Selective attention | 8 weeks
  The Stroop Task will be used to assess working memory at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment. The number of words, colors, and number of color words within a set time will be measured, as well as the number of errors. Larger amounts of errors reflect worse selective attention, whereas higher numbers of words, colors, and number of color words completed reflect better selective attention.
Inhibitory control - stop signal task | 8 weeks
  The Stop-signal task will be used to assess inhibitory control at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment.
Inhibitory control - reversal learning | 8 weeks
  A reversal learning task will be used to assess inhibitory control at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment.
Reward-based decision-making | 8 weeks
  A monetary delay-discounting task/questionnaires and the Balloon Analogue Risk task will be used to assess reward-based decision-making at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment. The primary outcome measures include the number of balloon pumps and earnings, with more pumps and earnings reflecting greater risk.
Resting state functional connectivity | 8 weeks
  Striatum resting state functional connectivity will be measured with a functional magnetic resonance imaging scan at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment.
Task-based brain activity (functional magnetic resonance imaging) - balloon analog risk | 8 weeks
  Performance on a cognitive task (the Balloon Analog Risk Task) will be assessed during a functional magnetic resonance imaging scan at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment.
Task-based brain activity (functional magnetic resonance imaging - stop signal | 8 weeks
  Performance on a cognitive task the (Stop Signal Task), will be assessed during a functional magnetic resonance imaging scan at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment.
Decision making under risk and ambiguity | 8 weeks
  A task involving decision making under during differing types of risk and ambiguity will be used to determine decision making under risk and ambiguity at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment. The Risk and Ambiguity Task measures tolerance for risk under conditions of known risk (alpha) and unknown risk (beta).
Loss Aversion | 8 weeks
  A computer task and written questionnaire assessing loss preferences will be used to assess loss aversion at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment.
Motor Function | 8 weeks
  A finger tapping test will be to assess motor function at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment. The number of finger taps in 10 seconds will be recorded three times per hand, and averaged to create the primary outcome measure reflecting motor function.

OTHER OUTCOMES:
Personality - impulsivity | 8 weeks
  Self-report of impulsivity will be measured at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment with the Barratt Impulsiveness Scale (11). The total score will be calculated as measured at both time points as the primary outcome measure.
Personality - novelty seeking | Baseline
  Self-report of novelty seeking will be measured at baseline prior to the EX or CON intervention using the Temperament and Character Inventory.
Personality - reward dependence | Baseline
  Self-report of reward dependence will be measured at baseline prior to the EX or CON intervention using the Temperament and Character Inventory.
Methamphetamine Craving | 8 weeks
  Self-report of craving of methamphetamine will be measured at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment using the Brief Meth Craving Scale. A total summary score is calculated and used as the primary outcome measure.
Cocaine Craving | 8 weeks
  Self-report of craving of cocaine will be measured at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment using the Cocaine Craving Questionnaire-Brief. A total summary score is calculated and used as the primary outcome measure.
Personality- risk taking | 8 weeks
  Self-report of risk perceptions and risk behaviors will be measured at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment using the Domain Specific Risk Taking Scale. Three scores will be computed: Risk Taking, Risk Perception, and Expected Benefits and changes in these scores will be measured at both time points.
Stimulant Withdrawal Score | 8 weeks
  Self-report of withdrawal symptoms from stimulants will be measured at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment using the Amphetamine Cessation Symptom Assessment. This 15 item questionnaire assesses acute (within the past 24 hours) craving, with lower scores reflecting lower craving. Changes in the total score will be assessed.
Smoking Withdrawal Score | 8 weeks
  Self-report of withdrawal symptoms from tobacco will be measured at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment using the Shiffman-Jarvik Withdrawal Scale on each scan day. This scale consists of 25 items assessing acute withdrawal, with lower scores reflecting lower withdrawal. Changes in the total score will be assessed.
Sleep Quality Rating | 8 weeks
  Self-report of sleep quality symptoms will be measured at baseline prior to exercise (EX) and after 8 weeks of EX (vs. CON) treatment using the Pittsburgh Sleep Quality Inventory. The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month.
State and trait anxiety | 8 weeks
  Self-report of anxiety symptoms will be measured at baseline prior to exercise (EX) and weekly during the 8 weeks of EX (vs. CON) treatment using the Speilberger State-Trait Anxiety Inventory.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT03709667/ICF_000.pdf